CLINICAL TRIAL: NCT03125694
Title: Efficacy, Durability, Safety, and Tolerability of Sitagliptin vs. Pioglitazone as add-on Treatments in Patients With Type 2 Diabetes Uncontrolled on the Full-dose Metformin Plus Sulfonylurea: a 52-week, Randomized, Open-label, Parallel-group, Phase 3 Clinical Trial
Brief Title: Sitagliptin vs. Pioglitazone as add-on Treatments in Patients With Type 2 Diabetes Uncontrolled on the Full-dose Metformin Plus Sulfonylurea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Esteghamati, Clinical Professor of Medicine, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9311160040
Record Dates: First submitted 2017-03-22; First posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Uncontrolled Type 2 Diabetes Mellitus
MeSH Terms: interventions — Sitagliptin Phosphate; Pioglitazone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sitagliptin (Active Comparator)
  Interventions: Drug: Sitagliptin 100mg
- Pioglitazone (Active Comparator)
  Interventions: Drug: Pioglitazone 30 mg

INTERVENTIONS:
Drug: Sitagliptin 100mg — Sitagliptin arm took sitagliptin 100 mg daily in combination with metformin 500 mg QID and gliclazide 80 mg TDS for 52 weeks
  Arms: Sitagliptin
Drug: Pioglitazone 30 mg — Pioglitazone arm took pioglitazone 30 mg daily in combination with metformin 500 mg QID and gliclazide 80 mg TDS for 52 weeks
  Arms: Pioglitazone

SUMMARY:
This study has been designed to investigate the comparative effects of sitagliptin vs. pioglitazone as add-on treatments in patients with type 2 diabetes who were uncontrolled on the full-dose of metformin and sulfonylurea

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes according to the American Diabetes Association
* Baseline level of 7% ≤ A1C < 11% despite a minimum 6 months period of active treatment with metformin 2000 mg/day plus gliclazide 240 mg/day (uncontrolled type 2 diabetes)

Exclusion Criteria:

* Acute or chronic diseases of heart, lung, kidney,
* Active or past infectious conditions
* Malignancy

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean glycated hemoglobin (A1C) levels by sitagliptin vs. pioglitazone | 52 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tehran University of Medical Sciences, Tehran, Iran